CLINICAL TRIAL: NCT04281810
Title: Effects of Transcutaneous Electrical Diaphragmatic Stimulation on Respiratory Function in Patients With Prolonged Mechanical Ventilation
Brief Title: Transcutaneous Electrical Diaphragmatic Stimulation in PMV Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 201700096A3D001
Record Dates: First submitted 2020-02-18; First posted 2020-02-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Mechanical Ventilation
Keywords: electrical stimulation; diaphragmatic; weaning; respiratory muscle

STUDY DESIGN:
Who Masked: Participant
Masking Description: Subjects were not informed of the results of allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEDS (Experimental): Subjects received transcutaneous electrical diaphragm stimulation (TEDS) for 30min/ day till the end of the weaning trial
  Interventions: Device: transcutaneous electric diaphragm stimulation
- Control (No Intervention): Subjects received similar medical treatment except for the TEDS program.

INTERVENTIONS:
Device: transcutaneous electric diaphragm stimulation — The electrodes were placed on the parasternal region beside the xiphoid process; and the sixth and seventh intercostal spaces in line with the mid-axillary line. TEDS was set as biphasic waves, frequency of 30 Hz, pulse width of 400 μs, and rise time of 0.7s.
  Arms: TEDS

SUMMARY:
Muscle atrophy and diaphragm dysfunction are common with prolonged mechanical ventilation (PMV). Electrical stimulation has been shown to be beneficial in severe chronic heart failure and chronic obstructive pulmonary disease. However, its effect on PMV is unclear. This study examined the effects of transcutaneous electrical diaphragmatic stimulation (TEDS) on respiratory muscle strength and weaning outcomes in patients with PMV.

DETAILED DESCRIPTION:
Patients on ventilation for ≥21 days were randomly assigned to TEDS and control groups. The TEDS group received muscle electrical stimulation for 30 min/session/day throughout the intervention. Weaning parameters (tidal volume, respiratory rate, and rapid shallow breathing index) and respiratory muscle strength (Pimax, Pemax) were assessed. The hospitalization outcome, including weaning rate and length of stay, was followed up until discharge.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years;
* MV for > 6 h/day for > 21 days;
* Medical stability (PaO2 ≥ 60 mmHg at 40% FiO2, absence of signs and symptoms of infection, and hemodynamic stability).

Exclusion Criteria:

* Acute lung or systemic infection, hemodynamic instability, patients with pacemakers, abdominal distention, and pregnancy.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2018-09-29 (Actual); Study Completion 2019-07-25 (Actual)

PRIMARY OUTCOMES:
tidal volume | 1st day of intervention
  The tidal volume was measured by a spirometer
tidal volume | through study completion,an average of 4 weeks
  The tidal volume was measured by a spirometer
rapid shallow breathing index | 1st day of intervention
  respiratory rate/tidal volume
rapid shallow breathing index | through study completion,an average of 4 weeks
  respiratory rate/tidal volume
respiratory muscle strength (maximal inspiratory pressure) | the 1st day of intervention
  pressure gauge
respiratory muscle strength (maximal expiratory pressure) | the 1st day of intervention
  pressure gauge
respiratory muscle strength (maximal inspiratory pressure) | through study completion,an average of 4 weeks
  pressure gauge
respiratory muscle strength (maximal expiratory pressure) | through study completion,an average of 4 weeks
  pressure gauge

SECONDARY OUTCOMES:
weaning rate | through study completion,an average of 7 weeks
  ventilator weaning results (weaning successful/failure)
length of stay in respiratory care center | through study completion,an average of 7 weeks
  the total days of stay in respiratory care center

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Fei Hsin, Principal Investigator — Chang Gung Memorial Hospital; Yen-Huey Chen, Study Director — Chang Gung University
Locations (1):
- Chang Gung University, Taoyuan, Tao-Yuan, Taiwan

IPD SHARING:
Plan to Share IPD: No